CLINICAL TRIAL: NCT03635320
Title: A Prospective Study Evaluating Trochanteric Fixation Nail Advanced (TFNA) in a Chinese Patient Population
Brief Title: The CHINA TFNA Study
Acronym: TFNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Synthes GmbH (Industry)
Collaborators: Johnson & Johnson Medical (Shanghai) Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DPS-201502; 2018l0002 (Other: CFDA)
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Results first posted 2021-05-21 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Femur Fractures
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Intervention Model Description: The study population will include 188 patients with proximal femur fracture undergoing internal fixation using an intramedullary nail.
  Subjects will be randomized in a 1:1 ratio to receive either the investigational TFNA devices (n=94) or to the control PFNA-II devices (n=94).
Who Masked: Participant
Masking Description: Only patient is masked during the study. He/she will be notified during inform consent that either treatment will be used but they will not be informed exactly which group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- investigational group (Experimental): using Trochanteric Fixation Nail Advanced to treat the fracture
  Interventions: Device: TFNA
- the control group (Active Comparator): Using Proximal Femoral Nail Antirotation to treat the fracture
  Interventions: Device: PFNA-II

INTERVENTIONS:
Device: TFNA — intramedullary nail 'Trochanteric Fixation Nail Advanced' to treat proximal femur fracture undergoing internal fixation
  Arms: investigational group
Device: PFNA-II — intramedullary nail ' Proximal Femoral Nail Antirotation' to treat proximal femur fracture undergoing internal fixation
  Arms: the control group

SUMMARY:
This is a prospective, multicenter, randomized, controlled, two-arm, non-inferiority study which will be conducted in China to support registration of a cephalomedullary nailing system (TFNA) that currently is available globally. The study will compare the safety and the effectiveness of two intramedullary nails (the investigational group is TFNA and the control group is PFNA-II).Patients enrolled at each site will be randomized in a ratio of 1:1, i.e. one patient assigned to surgery implanted with TFNA for each patient assigned to PFNA-II. Separate block randomization schedules within each site will be used to ensure equal distribution of treatment and control patients. Up to 15 centers will be approved to participate in this study.

Patient will be clinically followed after surgery at 1, 6, 12 and 24 weeks. The data up to and including 24 week follow up visit will be used in determining the primary safety and effectiveness of the TFNA.

The primary objective of this study is to evaluate whether fracture union rate, evaluated 24 weeks after proximal femur fracture, for the investigational TFNA intramedullary nail is non-inferior to that for currently available control product PFNA-II in patients with proximal femur fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patients with unilateral proximal femur fractures that will be treated with intramedullary nail internal fixation
3. According to AO fracture classification, subjects with following fracture type:

   1. Pertrochanteric (31-A1 and 31-A2)
   2. Intertrochanteric (31-A3)
   3. Trochanteric area (31-A1/A2/A3) with diaphyseal extension
4. Subject must be comfortable with speaking and understanding questions and responses in an available translated language for patient reported outcomes (PROs)

Exclusion Criteria:

1. Subject does not provide voluntary consent to participate in the study
2. The subject is a woman who is pregnant or lactating
3. Fractures where the operative treatment will occur more than three weeks after the primary injury
4. Patients with femoral head fractures and femoral neck fractures (AO classification 31-B and 31-C)
5. Pathological fracture (e.g., primary or metastatic tumor)
6. Serious soft tissue injury, judged by the investigator, will impact the union of the fracture, combined vascular injury, and combined osteofascial compartment syndrome
7. Multiple systemic injuries judged by researchers not suitable for enrollment, or orthopaedic fractures in other bones at three or more sites
8. Revision surgeries (for example, due to malunion, nonunion or infection)
9. Concurrent medical conditions judged by researchers not suitable for enrollment, such as: diabetes, metabolic bone disease, post-polio syndrome, poor bone quality, prior history of poor fracture healing, etc
10. Patients with anaesthetic and surgical contraindications
11. Patients known to be allergic to implant components
12. Patients who are currently using chemotherapeutics or accepting radiotherapy, use systematically corticosteroid hormone or growth factor, or long-term use sedative hypnotics (continuous use over 3 months) or non-steroidal anti-inflammatory drugs (continuous use over 3 months)
13. Intemperance judged by researchers not suitable for enrollment (e.g., excessive daily drinking or smoking, drug abuse);
14. Patients participated into other clinical trial in the previous 3 months;
15. Patients with bad compliance judged by researchers and cannot complete the test according to test scheme, such as schizophrenia and dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manyi Wang, Dr, Principal Investigator — Beijing Jishuitan Hospita; Vivian Li, Dr, Study Director — Johnson & Johnson Medical (Shanghai) Ltd.
Locations (9):
- China (9):
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - Peking University third Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical university, Guangzhou, Guangdong
  - University of Hong Kong shenzhen hospital, Shenzhen, Guangdong
  - The Second AffiliatedHospital of Zhejiang University of Medicine, Hangzhou, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Nantong
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Zhang L, Pan Z, Zheng X, Wang Q, Tang P, Zhou F, Liu F, Yu B, Leung FKL, Wu A, Hughson S, Chen Z, Blauth M, Rosner A, Sparks C, Wang M. Prospective randomized multicenter noninferiority clinical trial evaluating the use of TFN-advancedTM proximal femoral nailing system (TFNA) for the treatment of proximal femur fracture in a Chinese population. Eur J Trauma Emerg Surg. 2023 Jun;49(3):1561-1575. doi: 10.1007/s00068-023-02231-x. Epub 2023 Feb 13. PMID 36780014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred eighty-eight subjects were included in this study and randomly assigned to a study group; enrollment included 94 in the study group and 94 in the control group. Subjects were clinically followed after surgery at 1, 6, 12 and 24 weeks at the hospital.
Pre-assignment Details: Subjects required to meet inclustion/exclusion prior to receiving device. 4 subjects were screened but not randomized: 1 subject withdrew ICF before randomization, 1 subject didn't meet inclusion criteria 4, 1 subject met exclusion criteria 9 and 10, 1 subject met exclusion criteria 15.
Groups:
- TFNA Group (Study Group): intramedullary nail 'Trochanteric Fixation Nail Advanced' to treat proximal femur fracture undergoing internal fixation
- PFNA-II Group (Control Group): intramedullary nail 'Proximal Femoral Nail Antirotation' to treat proximal femur fracture undergoing internal fixation
Period: Overall Study
Arm/Group | TFNA Group (Study Group) | PFNA-II Group (Control Group)
Started (Participated in randomization) | 94 | 94
FAS (Full Analysis Set (FAS): The data set constituted by all subjects who participate in the randomized study and receive the product (implant).) | 93 (1 subject was not implanted the device) | 92 (2 subjects were not implant the device)
PPS (Per Protocol Set (PPS): A set of subjects that complete the trial, excluding those with serious protocol violation affecting the primary efficacy endpoints.) | 81 (11 subjects early discontinued and didn't complete the trial which were excluded from PPS, 1 subject had a risk of unblinding, which was excluded from the PPS.) | 83 (6 subjects early discontinued and didn't complete the trial which were excluded from PPS, 1 subject didn't undergo the evaluation or laboratory examination required by the clinical trial, 1 subject violated the inclusion/exclusion criteria and 1 subject used the device beyond the scope of the specifications, which were excluded from the PPS.)
Completed (Completed the study visits) | 82 | 86
Not Completed | 12 | 8
Not completed — not implanted the device | 1 | 2
Not completed — Withdrawal by Subject | 11 | 6

BASELINE CHARACTERISTICS:
Population: 3 subjects were not implanted with any device, so total 185 subjects were included in FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | TFNA Group (Study Group) | PFNA-II Group (Control Group) | Total
Number analyzed (Participants) | 93 | 92 | 185
Age, Continuous [Mean (Full Range); unit: Years] — Population: based on the FAS
  Years | 77.8 [30 to 91] | 74.1 [29 to 91] | 75.9 [29 to 91]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: based on the FAS
  Participants
    Female | 64 | 59 | 123
    Male | 29 | 33 | 62
Race/Ethnicity, Customized [Number; unit: Participants] — Population: based on the FAS
  Participants
    Han(Asian) | 89 | 91 | 180
    Others | 4 | 1 | 5
Medical history [Count of Participants; unit: Participants] — Population: based on the FAS
  Participants
    Osteoporosis: Yes | 56 | 55 | 111
    Osteoporosis: No | 37 | 37 | 74
    Malnutrition: Yes | 13 | 14 | 27
    Malnutrition: No | 80 | 78 | 158
    Anemia: Yes | 42 | 38 | 80
    Anemia: No | 51 | 54 | 105
    Hormone deficiency: Yes | 1 | 0 | 1
    Hormone deficiency: No | 92 | 92 | 184
    Diabetes: Yes | 28 | 18 | 46
    Diabetes: No | 65 | 74 | 139
    Smoke within one year: Yes | 5 | 5 | 10
    Smoke within one year: No | 88 | 87 | 175
    Drink within one year: Yes | 3 | 5 | 8
    Drink within one year: No | 90 | 87 | 177

OUTCOME MEASURES:

1. Primary Outcome: Successful Fracture Union Rate 24 Weeks After Surgery
Description: The number of achieving fracuture union at 24 weeks of each group will be counted and the percentage will be calculated.
  Fracture union success is a composite endpoint; in order for an individual subject's surgery implanted with TFNA or PFNA-II to be considered successful he/she must satisfy all of the following criteria:
  1. No focal tenderness or lengthwise percussion pain, or abnormal movement
  2. The frontal/lateral X-ray examination shows the vague or no fracture gap, or the continuous callus passing across the fracture line
  3. No deformation or breakage is found in the test product
Time Frame: 24 weeks
Population: based on PPS
Measure: Count of Participants; unit: Participants
Arm/Group | TFNA Group (Study Group) | PFNA-II Group (Control Group)
Number analyzed (Participants) | 81 | 83
Participants | 81 | 83
Statistical Analysis 1: Comparison: TFNA Group (Study Group) vs PFNA-II Group (Control Group); Test type: Non-Inferiority — non-inferiority margin of -10%; Newcombe-Wilson scoring method; Using the Newcombe-Wilson scoring method, the difference of fracture union rate between the TFNA group and the PFNA-II group was 0; 95%CI = 0, 95% CI 2-sided [-4.53 to 4.42] — If the lower limit of 95% CI of the difference in the rates of the study group and the control group is greater than the non-inferiority margin of -10%, then the investigational product is considered non-inferior to the control product

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were recorded starting at the time of subject randomization, until subject completion of study (24 weeks follow-up visit after surgery). All AEs were followed until the AE resolved, stabilized, or the study was completed.
Description: Judged the relationship between them and the products, and summarized the occurrence types of AEs for the safety evaluation of the product.
Arm/Group | TFNA Group (Study Group) | PFNA-II Group (Control Group)
All-Cause Mortality (participants affected / at risk) | 2/93 | 1/92
Serious Adverse Events (participants affected / at risk) | 18/93 | 16/92
Other Adverse Events (participants affected / at risk) | 93/93 | 89/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TFNA Group (Study Group) (N=93) | PFNA-II Group (Control Group) (N=92)
Device-related (Product Issues) | 0 (0) | 0 (0) — The Serious Adverse Events which was judged as Device-related Adverse Events
Non-device related (Product Issues) | 18 (22) | 16 (21) — The Serious Adverse Events which was judged as Non-device related Adverse Events
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TFNA Group (Study Group) (N=93) | PFNA-II Group (Control Group) (N=92)
Device related (Product Issues) | 0 (0) | 0 (0) — The Adverse Events which was judged as Device-related Adverse Events
Non-device related (Product Issues) | 93 (362) | 89 (361) — The Serious Adverse Events which was judged as Non-device related Adverse Events

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal investigator and institution will not be able to publish single-center study data until combined results of the multicenter study are published. If multicenter publication is not performed within 12 months after the end or if sponsor notifies principal investigator and institution in writing that the multicenter study results will not be published, the principal investigator and institution may publish the results of their studies separately in accordance with contract.

DOCUMENTS (2):
  • Study Protocol (2019-01-08): https://cdn.clinicaltrials.gov/large-docs/20/NCT03635320/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT03635320/SAP_001.pdf